CLINICAL TRIAL: NCT03602768
Title: Evaluation of Online Cognitive Fitness Programs
Brief Title: Evaluation of the Online Memory & Aging Program and Online Goal Management Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Collaborators: Centre for Aging and Brain Health Innovation (Other)
Responsible Party: Principal Investigator, Brian Levine, Senior Scientist, Baycrest
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17-24
Record Dates: First submitted 2018-07-12; First posted 2018-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Aging; Cognitive Decline
Keywords: Healthy aging; executive functions; memory; cognitive training; cognitive intervention; subjective cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants are screened, undergo a battery of cognitive testing for the pre-test, and then are randomly assigned to one of four intervention groups: MAP, GMT, Cambridge Brain Sciences brain training (active control), or waitlist. After intervention, the participants take the same test battery and complete it once more at 6 week followup.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study personnel who conduct screening and send pre/post-test surveys to participants are all blinded.
  Randomizer is blinded to all participant pre-test outcomes. Care providers know what their participants are doing, but not aware of the full study design, including details of the other conditions or outcome test characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Goal Management Training (Experimental): The online version of GMT with a therapist on the back-end monitoring progress and giving feedback throughout the program. Online GMT takes 5-9 weeks (self-paced) to complete 9 modules involving instructional video with interactive content, practice of cognitive strategies through games, and between-module exercises.
  Interventions: Behavioral: Goal Management Training
- Memory & Aging Program (Experimental): The online version of MAP with a therapist moderator on the course discussion pages. MAP takes 5-9 weeks (self-paced) to complete 8 modules involving instructional video with interactive content and practice of memory strategies through various exercises.
  Interventions: Behavioral: Memory & Aging Program
- Cambridge Brain Sciences Training (Placebo Comparator): This is a commercial and research brain training platform, composed of 7 games that are online adaptations of the standard measures of cognition including working memory and spacial planning.
  Interventions: Behavioral: Cambridge Brain Sciences
- Waitlist (No Intervention): Participants randomized to this arm will receive no additional information or access to intervention programs until after the follow up testing measures are collected, at which point they will be given access to the intervention of their choosing.

INTERVENTIONS:
Behavioral: Goal Management Training — Pre-recorded videos and games combine psycho-education, targeted skills training, and mindfulness practice to teach a system where participants can take control of their attention and cognitive faculties.
  Other Names: GMT
  Arms: Goal Management Training
Behavioral: Memory & Aging Program — Pre-recorded videos and activities combine psycho-education, memory strategy training, and social support to educate about normal memory change in aging, normalize the experience of participants going through it, and equip them to handle age-related memory change.
  Other Names: MAP
  Arms: Memory & Aging Program
Behavioral: Cambridge Brain Sciences — Commercial brain training software available for subscription to the general public and for research studies.
  Arms: Cambridge Brain Sciences Training

SUMMARY:
The current study is designed to test the effectiveness of online programs for memory and executive functions in healthy aging. The investigators are testing online adaptations of two cognitive interventions that have been extensively studied, validated, and implemented in clinical settings: The Memory & Aging Program (MAP) targets normal memory change in healthy aging, and Goal Management Training (GMT) targets executive functioning deficits in a variety of cognitive and neurological conditions including healthy aging. Both programs combine psycho-education, targeted skills training and clinical support to empower participants with knowledge and strategies to harness their cognitive faculties. These programs are being tested against a waitlist control as well as against a commercial/research brain training platform (Cambridge Brain Sciences) in a design comparing performance on memory and executive functioning measures before and after the interventions/controls. The main hypothesis is that MAP will lead to memory-specific improvements above control conditions, whereas GMT will lead to greater improvements in measures of executive functions relative to controls.

ELIGIBILITY:
Inclusion Criteria:

* Available to participate in all testing and intervention sessions and access to a computer
* Computer familiarity
* Cognitive complaint/concern/frustration

Exclusion Criteria:

* Health conditions with major effects on cognition, including a current or previous history of stroke, brain surgery, or diagnosed neurological disorder;
* Dependence in instrumental activities of daily living
* Cognitive impairment, defined as performance below cutoff for cognitive impairment on a standardized cognitive screening measure, the modified Telephone Interview for Cognitive Status (Welsh et al., 1993)
* Affective impairment, defined as performance below cutoff for depression on standardized depression screen, the PHQ 2/9 (Yesavage et al., 1983)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Change in dysexecutive functioning | Pre-intervention; immediate post-intervention; 6 weeks following intervention completion.
  Dysexecutive Functioning Index (DEX) questionnaire measures self-reported deficits in executive functions, and is composed of one scale with scores ranging from 0-80, where higher scores indicate greater executive deficit.
Change in cognitive failures | Pre-intervention; immediate post-intervention; 6 weeks following intervention completion.
  Cognitive Failures Questionnaire (CFQ) measures self-reported failures in perception, memory, and motor function. It contains a single scale with scores ranging from 0-100, where higher scores indicate greater degree of impairment.
Change in memory knowledge score | Pre-intervention (post-randomization); immediate post-intervention; 6 weeks following intervention completion.
  Memory Knowledge Quiz quantifies memory, lifestyle, and strategy knowledge. It is scored from 0-25, with higher scores indicating more knowledge about knowledge of lifestyle factors affecting memory and strategies to remember.
Change in memory strategy toolbox use | Pre-intervention; immediate post-intervention; 6 weeks following intervention completion.
  Memory Strategy Toolbox quantifies application of strategies in memory-demanding everyday situations. It is scored from 0 - 6, with higher scores indicating increased ability to apply memory strategy toolbox.
Change in Multifactorial Metamemory Questionnaire (MMQ) | Pre-intervention; immediate post-intervention; 6 weeks following intervention completion.
  Quantifies subjective memory abilities, satisfaction, and strategy use. The MMQ contains 3 sub scales, but we are using total score as our outcome variable. MMQ total scores range from 0 - 228, with higher scores indicting high self-reported memory performance, satisfaction with it, and use of memory strategies.

SECONDARY OUTCOMES:
Change in Patient-Specific Functional Scale | Pre-intervention (post-randomization); immediate post-intervention; 6 weeks following intervention completion.
  Quantifies the impact of memory changes on daily activities and self-image. Is scored from 0 -10, with higher scores indicating greater ability to perform function, and taken as an average across number of activities scored.
Change in Impact of Memory Change on Daily Activities | Pre-intervention (post-randomization); immediate post-intervention; 6 weeks following intervention completion.
  Memory Impact Questionnaire (MIQ) quantifies the impact of memory changes on daily activities and self-image. The MIQ has three sub scales: Lifestyle Restriction, Positive Coping and Negative Emotion, and total score will be used as the outcome variable. Scores range from 0 - 204, with higher scores indicating greater impact of memory change on daily activities and self image.
Change in intentions to seek medical attention | Pre-intervention (post-randomization); immediate post-intervention; 6 weeks following intervention completion.
  Quantifies change in intentions to seek medical attention pertaining to memory concerns.
Change in Cambridge Brain Sciences online cognitive assessment | Pre-intervention (post-randomization); immediate post-intervention; 6 weeks following intervention completion.
  Battery of tasks that assess aspects of memory and reasoning.
Change in associative memory | Pre-intervention (post-randomization); immediate post-intervention; 6 weeks following intervention completion.
  Face-name task tests associative memory and sensitivity (d') will be measured as the outcome score.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Levine, PhD, Principal Investigator — Rotman Research Institute
Locations (1):
- Baycrest Health Sciences, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brandt, J., Spencer, M., & Folstein, M. (1988). The Telephone Interview for Cognitive Status. Neuropsychiatry, Neuropsychology, & Behavioral Neurology, 1(2), 111-117.
- [Background] Broadbent DE, Cooper PF, FitzGerald P, Parkes KR. The Cognitive Failures Questionnaire (CFQ) and its correlates. Br J Clin Psychol. 1982 Feb;21(1):1-16. doi: 10.1111/j.2044-8260.1982.tb01421.x. PMID 7126941
- [Background] Burgess, P. W., Alderman, N., Wilson, B. A., Evans, J. J., & Emslie, H. (1996). The dysexecutive questionnaire. Behavioural assessment of the dysexecutive syndrome. Bury St. Edmunds, UK: Thames Valley Test Company.
- [Background] Hampshire A, Highfield RR, Parkin BL, Owen AM. Fractionating human intelligence. Neuron. 2012 Dec 20;76(6):1225-37. doi: 10.1016/j.neuron.2012.06.022. PMID 23259956
- [Background] Levine B, Stuss DT, Winocur G, Binns MA, Fahy L, Mandic M, Bridges K, Robertson IH. Cognitive rehabilitation in the elderly: effects on strategic behavior in relation to goal management. J Int Neuropsychol Soc. 2007 Jan;13(1):143-52. doi: 10.1017/S1355617707070178. PMID 17166313
- [Background] Levine B, Robertson IH, Clare L, Carter G, Hong J, Wilson BA, Duncan J, Stuss DT. Rehabilitation of executive functioning: an experimental-clinical validation of goal management training. J Int Neuropsychol Soc. 2000 Mar;6(3):299-312. doi: 10.1017/s1355617700633052. PMID 10824502
- [Background] Levine B, Schweizer TA, O'Connor C, Turner G, Gillingham S, Stuss DT, Manly T, Robertson IH. Rehabilitation of executive functioning in patients with frontal lobe brain damage with goal management training. Front Hum Neurosci. 2011 Feb 17;5:9. doi: 10.3389/fnhum.2011.00009. eCollection 2011. PMID 21369362
- [Background] Troyer, A. K. (2001). Improving memory knowledge, satisfaction, and functioning via an education and intervention program for older adults. Aging, Neuropsychology, and Cognition, 8(4), 256-268
- [Background] Troyer AK, Murphy KJ, Anderson ND, Moscovitch M, Craik FI. Changing everyday memory behaviour in amnestic mild cognitive impairment: a randomised controlled trial. Neuropsychol Rehabil. 2008 Jan;18(1):65-88. doi: 10.1080/09602010701409684. PMID 17943615
- [Background] Troyer AK, Rich JB. Psychometric properties of a new metamemory questionnaire for older adults. J Gerontol B Psychol Sci Soc Sci. 2002 Jan;57(1):P19-27. doi: 10.1093/geronb/57.1.p19. PMID 11773220
- [Background] Walker SN, Sechrist KR, Pender NJ. The Health-Promoting Lifestyle Profile: development and psychometric characteristics. Nurs Res. 1987 Mar-Apr;36(2):76-81. PMID 3644262
- [Background] Welsh, K. A., Breitner, J.C.S., & Magruder-Habib, K.M. (1993) Detection of dementia in the elderly using telephone screening of cognitive status. Neuropsychiatry, Neuropsychology, and Behavioral Neurology, 6, 103-110.
- [Background] Wiegand MA, Troyer AK, Gojmerac C, Murphy KJ. Facilitating change in health-related behaviors and intentions: a randomized controlled trial of a multidimensional memory program for older adults. Aging Ment Health. 2013;17(7):806-15. doi: 10.1080/13607863.2013.789000. Epub 2013 Apr 23. PMID 23611105
- [Derived] Yusupov Rose I, Lass JW, D'Amico D, Zhu L, Rich JB, Levine B, Vandermorris S, Troyer AK. A self-guided e-learning program improves metamemory outcomes in healthy older adults: a randomized controlled trial. Aging Ment Health. 2025 Jun;29(6):1090-1099. doi: 10.1080/13607863.2024.2438839. Epub 2024 Dec 13. PMID 39672101

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT03602768/Prot_SAP_ICF_000.pdf